CLINICAL TRIAL: NCT02853175
Title: Diagnostic Accuracy of Lung MRI to Detect Allergic Broncho-pulmonary Aspergillosis in Cystic Fibrosis
Brief Title: Lung MRI and Allergic Broncho-pulmonary Aspergillosis in Cystic Fibrosis
Acronym: MRAB
Status: Completed | Type: Observational
Sponsor: Hôpital Haut Lévêque (Other)
Collaborators: University Hospital, Bordeaux (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor-Investigator, Hôpital Haut Lévêque, MD-PhD, Hôpital Haut-Lévêque
Organization: Hôpital Haut-Lévêque (Other)
Other Study IDs: ANR-10-LABX-57
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Cystic Fibrosis; ABPA
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with both CF and ABPA: Patients with both cystic fibrosis and allergic broncho-pulmonary aspergillosis (ABPA).
  The diagnosis of ABPA (Gold Standard) rely on routine dosage of total immunoglobulin E (IgE), specific to Aspergillus IgE, specific to aspergillus Immunoglobulin G, eosinophilia on blood cell count, and imaging (infiltrate, mucoid impaction, central bronchiectasis)
- Patients with CF and no ABPA: Patients with both cystic fibrosis and no allergic broncho-pulmonary aspergillosis (ABPA).
  The diagnosis of ABPA (Gold Standard) rely on routine dosage of total immunoglobulin E (IgE), specific to Aspergillus IgE, specific to aspergillus Immunoglobulin G, eosinophilia on blood cell count, and imaging (infiltrate, mucoid impaction, central bronchiectasis)

SUMMARY:
In this diagnostic study, the aim is at evaluating the diagnostic accuracy of MRI (Magnetic Resonance Imaging) to detect allergic broncho-pulmonary aspergillosis in patients with cystic fibrosis.

DETAILED DESCRIPTION:
Allergic broncho-pulmonary aspergillosis (ABPA) is not rare in the context of cystic fibrosis (CF), with a prevalence reported between 2% to 16%. This complication is a diagnostic challenge for clinicians, since it is related with poorer outcome and higher worsening of the disease. Therefore, the treatment relies on corticosteroid and antifungal therapy and thus, it is important to detect with good sensitivity because CF patients are usually treated with antibiotics. However, the treatment is often difficult to be initiated because of potential secondary side effects related to diabetes mellitus, growth impairment, bone mineralisation or immunodepression. Therefore, there is a need for specific diagnostic tool to discriminate ABPA amongst other polymicrobial infection.

Lung MRI is a radiation-free imaging modality which offers the potential to combine several contrasts, in order to enable in vivo tissue characterization non-invasively. Investigators hypothesize that characterization of mucoid impaction using lung MR T1-weighted and T2-weighted contrasts may be a specific tool to diagnose ABPA in CF non invasively. Additional information on functional information related to ventilation and/or perfusion will be assessed using functional MR sequences, to assess the severity of small airway impairment. Moreover, the diagnostic value of structural alterations such as bronchiectasis, mucoid impaction and consolidation/atelectasis using either MRI with ultrashort echo times or CT using reduction of doses down to chest radiograph levels will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis proven by sweat chloride and genetic tests
* Age superior or equal to 6 year-old
* Diagnosis of ABPA available on the basis of the criteria by Cystic Fibrosis Foundation Consensus Conference
* No contraindication to perform MRI

Non-Inclusion Criteria:

. Age inferior to 6-year-old

* Cystic fibrosis not proven
* ABPA status not documented
* MRI contraindications: Pregancy, Magnetically activated implanted devices (cardiac pacemakers, insulin pumps, neurostimulators, cochlear implants...), metal inside the eye or the brain (aneurysm clip, ocular foreign body not compatible with MRI), cardiac valvular prothesis not compatible with MRI, subject with claustrophobia.

Exclusion Criteria: None

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients routinely followed-up for cystic fibrosis from chilhood to adulthood.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2014-01; Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of lung MRI for ABPA in CF owing to increased T1 and decreased T2 signal intensity of mucus | From date of inclusion until the date of final ABPA status diagnosis, assessed up to 12 months
  Measurement of sensitivity, specificity, positive predictive value, negative predictive value of lung MRI to diagnose ABPA in CF, owing to the presence of central mucoid impactions that appear both hyperintense on T1-weighted sequence and hypointense on T2-weighted sequence

SECONDARY OUTCOMES:
Diagnostic accuracy of quantitative measurement of central mucoid impaction signal on T1-weighted sequence and T2-weighted sequence | From date of inclusion until the date of final ABPA status diagnosis, assessed up to 12 months
  Measurement of sensitivity, specificity, positive predictive value, negative predictive value of lung MRI to diagnose ABPA in CF, owing to the quantitative measurement of signal from central mucoid impaction using T1-weighted and T2-weighted sequences
Diagnostic accuracy of hyperattenuated central mucoid impaction on chest computed tomography (CT) to detect ABPA in CF, using reduction of doses down to chest radiograph level | From date of inclusion until the date of final ABPA status diagnosis, assessed up to 12 months
  Measurement of sensitivity, specificity, positive predictive value, negative predictive value of lung MRI to diagnose ABPA in CF, owing to the presence of central mucoid impactions that appear hyperattenuated on chest CT
Diagnostic follow-up of patients ABPA status 1 year | From date of inclusion until the date of final ABPA status diagnosis, assessed up to 12 months
  Re-evaluation of diagnostic criteria for ABPA with up to 1-year follow-up in patients with undetermined ABPA status at initial evaluation
Diagnostic accuracy of MRI to detect ABPA in CF using various ABPA classifications | From date of inclusion until the date of final ABPA status diagnosis, assessed up to 12 months
  To assess the accuracy of lung MRI to detect ABPA in a CF patient cohort if various ABPA classification are used
Reproducibility of qualitative and quantitative imaging evaluations | From date of inclusion until the date of final ABPA status diagnosis, assessed up to 12 months
  To assess the intra-observer and inter-observer reproducibility of 2 readers to diagnose ABPA in CF using lung MRI
Diagnostic accuracy of morphological imaging using MRI with ultrashort echotimes | From date of inclusion until the date of final ABPA status diagnosis, assessed up to 12 months
  Measurement of sensitivity, specificity, positive predictive value, negative predictive value of lung MRI to diagnose ABPA in CF, owing to the presence of structural alterations
Diagnostic accuracy of morphological imaging using CT with reduction of doses down to chest radiograph level | From date of inclusion until the date of final ABPA status diagnosis, assessed up to 12 months
  Measurement of sensitivity, specificity, positive predictive value, negative predictive value of CT to diagnose ABPA in CF, owing to the presence of structural alterations
Reproducibility between MRI and CT with reduction of doses down to chest radiograph level to assess structural alterations | From date of inclusion until the date of final ABPA status diagnosis, assessed up to 12 months
  Measurement of agreement and concordance between MRI with ultrashort echo times and CT with reduction of doses down to chest radiograph level to assess the Bhalla score
Severity of small airway and perfusion alterations using functional MR sequences | From date of inclusion until the date of final ABPA status diagnosis, assessed up to 12 months
  Measurement of correlations between functional MRI and disease severity
Follow-up of disease severity under treatement | From date of inclusion until the date of final treatment, assessed up to 12 months
  Measurement of variation of MR outcomes under CF treatments

CONTACTS AND LOCATIONS:
Overall Officials: François Laurent, MD, Study Director — University Bordeaux Hospital
Locations (1):
- University Hospital Bordeaux, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No